CLINICAL TRIAL: NCT02100956
Title: Efficacy of Intrathecal Oxytocin in Patients With Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cessation of funding period prior to completion, due to slow recruitment during the pandemic
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00027272
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-11

CONDITIONS: Neuropathic Pain
Keywords: chronic pain; neuropathic pain
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Oxytocin, then Placebo (Experimental): The subject first received oxytocin 100 micrograms administered intrathecally (IT). After at least one week, they received normal saline placebo IT.
  Interventions: Drug: oxytocin 100 micrograms; Drug: Normal Saline (preservative free)
- Placebo, then Oxytocin (Experimental): The subject first received normal saline placebo intrathecally (IT). After at least one week, they then received oxytocin 100 micrograms administered IT.
  Interventions: Drug: oxytocin 100 micrograms; Drug: Normal Saline (preservative free)

INTERVENTIONS:
Drug: oxytocin 100 micrograms — oxytocin 100 micrograms administered intrathecally (IT)
Drug: Normal Saline (preservative free) — Normal Saline (preservative free) administered intrathecally (IT)

SUMMARY:
The purpose of the study is to determine the effect of oxytocin given into the spinal fluid on pain and areas and intensity of hyperalgesia and allodynia in patients with chronic neuropathic pain.

DETAILED DESCRIPTION:
Rationale: The investigators anticipate that oxytocin will be effective after spinal injection in humans to acutely relieve chronic neuropathic pain.

Objectives: Determine the effect of intrathecal oxytocin on pain and areas and intensity of hyperalgesia and allodynia in patients with chronic neuropathic pain.

Interventions: A computer generated randomization will be used to determine the group for each subject. Subjects will be randomized to receive an intrathecal injection of saline (placebo) or oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Weight < or equal to 240 pounds
* Neuropathic pain for > 6 months: with primary pain area below the umbilicus

Exclusion Criteria:

* Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug or lidocaine
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
* Pregnancy
* spinal cord stimulators, chronic intrathecal drug therapy, or oral opioid treatment for > 3 months at a current dose of > 100 milligram (mg) morphine per day or equivalent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06-19 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Eisenach JC, Curry RS, Houle TT. Preliminary results from a randomized, controlled, cross-over trial of intrathecal oxytocin for neuropathic pain. Pain Med. 2023 Sep 1;24(9):1058-1065. doi: 10.1093/pm/pnad051. PMID 37084261

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were not randomized, one because of an abnormal electrocardiogram and the other for lack of spontaneous neuropathic pain at rest. Six subjects were randomized and received the first intrathecal injection. Participant flow section includes randomized subjects only.
Period: First Injection
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: At Least One Week Between Injections
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Injection
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [41 to 52] | 54 [46 to 56] | 52 [40 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Visual Analog Scale Pain [Median (Inter-Quartile Range); unit: units on a scale] — The participant was asked to rate the level of their spontaneous current pain in the area of their neuropathic pain. They did so by drawing a vertical mark on a 10 cm horizontal line without gradations. Scale ranges from 0-10 with 0 meaning "No Pain" on the left end and 10 meaning "Worst Imaginable Pain" on the right end. The score is the number of cm of the mark from the left end of the horizontal line.
  units on a scale | 4.2 [3.9 to 6.2] | 2.6 [2.3 to 4.9] | 3.9 [2.8 to 6.4]

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Pain From Their Neuropathic Pain Disease
Description: Pain will be measured by visual analog scale, a 10 cm line with 0/"no pain" on the left end and 10/"pain as worse as can be" on the right end. The subject places a mark on the line and the score is determined by the distance in cm from the "no pain" end.
Time Frame: 240 minutes post injection
Population: The intention to treat population was defined as individuals who were randomized and received intrathecal drug on both study days of the trial. This includes subjects who completed both injections.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Oxytocin Injection: Participants who received intrathecal oxytocin injection on either the first or second study day
- Placebo Injection: Patients who received normal saline placebo injection on either the first or second study day.
Arm/Group | Oxytocin Injection | Placebo Injection
Number analyzed (Participants) | 5 | 5
score on a scale | 1.67 (0.87) | 2.43 (0.89)
Statistical Analysis 1: Comparison: Oxytocin Injection vs Placebo Injection; Null hypothesis was that there was no difference in VAS pain scale scores after intrathecal study drug injection between oxytocin and placebo. To account for repeated measures across time and drug conditions, VAS apin scale scores were analyzed using a linear mixed-effects model with random intercepts at the level of participant. Each outcome was regressed on fixed-effects for order of study day, study drug, time after injection, and drug x time interaction; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 6 months after second intrathecal injection, up to 6.5 months
Description: Peripheral oxyhemoglobin saturation, blood pressure, and heart rate were measured non invasively and recorded before and 15, 30, 60, 120, 180, 240, minutes after intrathecal injection. The electrocardiogram was continuously monitored. A neurologic examination was performed at intervals until 24 hours after injection. Serum sodium was assayed 24 hr after injection. Subjects were called 2, 3, 4, 5, 7 days, then weekly until one month and then at 6 months after the second intrathecal injection.
Arm/Group | Oxytocin Injection | Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin Injection (N=6) | Placebo Injection (N=6)
Post dural puncture headache (Nervous system disorders) | 0 (0) | 1 (1) — Subject developed a post dural puncture headache after the first intrathecal injection, beginning within 24 hr and lasting 5 days. It was treated with non-prescription analgesics and resolved spontaneously

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow recruitment and lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02100956/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02100956/ICF_000.pdf